CLINICAL TRIAL: NCT01251341
Title: Mechanisms of Meditation
Brief Title: The Compassion and Attention Longitudinal Meditation Study
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01AT004698 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Immune System Processes; Inflammatory Activation and Modulation; ANS Function
Keywords: inflammation; immune system; cytokines; meditation; compassion; attention
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Compassion Meditation Group (Experimental)
  Interventions: Behavioral: Cognitive-Based Compassion Training
- Health Education and Wellness Group (Active Comparator)
  Interventions: Behavioral: Adult Health Education Curriculum
- Mindful Attention Training (Experimental)
  Interventions: Behavioral: Mindful Attention Training

INTERVENTIONS:
Behavioral: Cognitive-Based Compassion Training — Eight-week training in compassion meditation, using a protocol developed by Geshe Lobsang Negi, Ph.D. of Emory University
  Arms: Compassion Meditation Group
Behavioral: Mindful Attention Training — Eight week training in mindful attention, using a protocol developed by B. Alan Wallace, Ph.D.
  Arms: Mindful Attention Training
Behavioral: Adult Health Education Curriculum — Eight week training in health and wellness, using a curriculum developed specifically for this study.
  Arms: Health Education and Wellness Group

SUMMARY:
The increasingly widespread use of meditation for stress-related emotional and medical conditions highlights the urgent need to rigorously evaluate mechanisms through which the benefits of practice might be conferred. Primary challenges in this regard include evaluating dose response relationships between practice time and outcomes; clarifying whether physiological and behavioral effects of meditation derive primarily from non-specific aspects of training or result from specific meditation practices; and identifying molecular mechanisms by which meditation might affect physiological responses relevant to stress-related illness. Recent findings from a cross-sectional study by our group indicate that young adults who are randomized to, and practice, compassion meditation demonstrate reduced inflammatory responses, less emotional distress, and reduced autonomic responses to a standardized laboratory psychosocial stressor (Trier Social Stress Test [TSST]) when compared to subjects randomized to an active control condition. However, as a result of the cross-sectional study design and lack of a meditation comparator arm, these results provide only partial insight into key issues outlined above regarding the role played by specific meditation procedures and/or practice time in observed physiological and behavioral outcomes. The primary hypothesis of the proposed work is that practicing a meditation procedure specifically designed to enhance empathic concern for others (i.e. compassion meditation) will optimize autonomic reactivity to psychosocial stress in a manner that results in diminished activation of peripheral inflammatory signaling pathways and reduced behavioral distress.

ELIGIBILITY:
Inclusion Criteria:

* Good medical health

Exclusion Criteria:

* current major depression
* current substance abuse
* lifetime history of schizophrenia or bipolar disorder type I as assessed by the Structured Diagnostic Interview for DSM-IV (SCID)
* suicidal ideation or suicide attempt within one year of study enrollment
* diagnosis of any serious ongoing medical condition including malignancy, auto-immune disease (i.e. rheumatoid arthritis, multiple sclerosis, Crohn's disease), cardiovascular disease (other than hypertension), seizure disorder, endocrinopathy, chronic infection (i.e. human immunodeficiency virus, hepatitis B or C), renal or hepatic insufficiency, or any other current or past medical or psychiatric condition that might increase the risk of study participation in the opinion of study personnel
* treatment with psychotropic medications within the last year (i.e. antidepressants, anxiolytics, psychostimulants or mood stabilizers)
* active ongoing psychiatric treatment at the time of enrollment.
* use of any psychotropic medication (i.e. antidepressants, anxiolytics, psychostimulants or mood stabilizers) within one year of screening.
* chronic use of anti-inflammatory/immunosuppressive agents, including, but not limited to, aspirin, non-steroidal anti-inflammatory agents, COX-2 inhibitors, corticosteroids, etanercept, infliximab, adalimumab or methotrexate.
* any significant past meditation training/experience (defined as meditating more than 3 times a week for a period longer than a month)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effects of compassion meditation on inflammatory and behavioral responses to psychosocial stress using a longitudinal design. | Five years
  Innate immune cytokine responses will be assessed before and after a psychosocial stressor to evaluate the differential impact of the two interventions and the active control.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona; Lobsang Tenzin Negi, PhD, Study Director — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States